CLINICAL TRIAL: NCT00566098
Title: Adoptive Immunotherapy Utilizing Activated Marrow Infiltrating Lymphocytes in the Autologous Transplant Setting in Multiple Myeloma
Brief Title: Activated White Blood Cells With ASCT for Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0770; P30CA006973 (NIH); NA_00012038 (Other: JHMIRB)
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — N(1)-methyl-2-lysergic acid diethylamide; Melphalan; Heptavalent Pneumococcal Conjugate Vaccine

ARMS (1):
- ASCT+MILs (Experimental): Autologous stem cell transplant with a conditioning regimen of melphalan 100 mg/m^2 on each of Days -2 and -1. Infusion of activated marrow infiltrating lymphocytes (MILs) on Day 3. PCV13 vaccine will be given before and/or after Day 0 depending on when participants are enrolled.
  Interventions: Biological: MILs; Drug: Melphalan; Biological: PCV13

INTERVENTIONS:
Biological: MILs
  Other Names: Marrow infiltrating lymphocytes; Activated marrow infiltrating lymphocytes; aMILs
Drug: Melphalan
  Other Names: Alkeran
Biological: PCV13
  Other Names: Prevnar

SUMMARY:
RATIONALE: Activating white blood cells in the laboratory may help them kill more cancer cells when they are put back in the body. This may be an effective treatment for patients undergoing a stem cell transplant for multiple myeloma.

PURPOSE: This phase I/II trial is studying the side effects of activated white blood cells and to see how well they work in treating patients who are undergoing a stem cell transplant for newly diagnosed stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and response rate of activated marrow infiltrating lymphocytes (aMILs) in patients undergoing autologous peripheral blood stem cell transplantation for newly diagnosed, stage II-III multiple myeloma.
* Determine the overall in vitro fold-expansion and assess pre- and post-expansion for myeloma T-cell specificity in assessing the feasibility of generating aMILs from myeloma patients.
* Assess the toxicity of aMILs.
* Evaluate the effect of aMILs on hematopoietic engraftment, including neutrophil engraftment, platelet engraftment, and primary graft failure (if failure occurs).
* Evaluate response rates utilizing the Blade criteria, including the complete response (CR) rate, near complete response (nCR) rate, very good partial response (VGPR) rate, partial response (PR) rate, minimal response (MR) rate, and overall response rate (CR, VGPR, PR, MR).

Secondary

* Evaluate T-cell reconstitution, including absolute lymphocyte counts, CD3+, CD4+, and CD8+ T-cell counts.
* Evaluate progression-free survival and overall survival.
* Evaluate anti-tumor immune response.
* Determine pneumococcal-specific vaccine responses.
* Determine delayed-type hypersensitivity (DTH) responses.

OUTLINE: Patients undergo collection of marrow infiltrating lymphocytes (MILs)* either at diagnosis prior to the initiation of induction therapy or upon completion of induction therapy. The MILs bone marrow product undergo ex vivo activation and expansion of T cells for 7-8 days to produce activated marrow infiltrating lymphocytes (aMILs). Patients then undergo stem cell mobilization and leukapheresis to collect the peripheral blood stem cells 12 days after mobilization. Patients receive melphalan IV over 20-30 minutes on days -2 and -1 and undergo a peripheral blood stem cell transplantation on day 0 as planned. Patients receive aMILs infusion on day 3. Patients receive pneumococcal polyvalent vaccine on day 21.

NOTE: *Patients who have completed induction therapy receive pneumococcal polyvalent vaccine approximately 2 weeks prior to MILs collection; patients undergoing MILs collection prior to starting induction therapy do not receive a pre-transplantation vaccine.

Blood and bone marrow samples are collected periodically for laboratory correlative studies.

After completion of study treatment, patients are followed periodically for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Newly diagnosed disease
  * Durie-Salmon stage II or III disease
* Measurable disease, defined by any of the following:

  * Measurable serum and/or urine M-protein levels documented and available prior to induction therapy
  * Positive serum free light chain assay
* Must have completed a minimum of 3 courses of myeloma specific therapy
* Candidate for autologous stem cell transplantation
* Patients who have achieved a complete remission at the time of bone marrow harvest for marrow infiltrating lymphocytes (MILs) expansion are not eligible
* No evidence of spinal cord compression
* Diagnosis of the following cancers are not allowed:

  * POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes)
  * Non-secretory myeloma (no measurable protein on serum free light chain assay)
  * Plasma cell leukemia
* No amyloidosis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and up to day 180
* Corrected serum calcium < 11 mg/dL and no evidence of symptomatic hypercalcemia
* Total bilirubin ≤ 2.0 times upper limit of normal (ULN)
* ALT ≤ 2.0 times ULN
* Serum creatinine < 2.0 mg/dL
* No history of other malignancy within the past 5 years, except adequately treated basal cell or squamous cell skin cancer
* No history of autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus) requiring systemic treatment

  * Hypothyroidism without evidence of Graves' disease or Hashimoto thyroiditis is allowed
* No infection requiring treatment with antibiotics, antifungal, or antiviral agents within the past 7 days
* No HIV infection
* No major organ system dysfunction including, but not limited to, the following:

  * New York Heart Association class III or IV congestive heart failure
  * Pulmonary disease requiring the use of inhaled steroids or bronchodilators
  * Renal, hepatic, gastrointestinal, neurologic, or psychiatric dysfunction that would impair ability to participate in the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hematopoietic stem cell transplantation
* At least 3 weeks since prior corticosteroids (i.e., glucocorticoids)
* At least 3 weeks since prior myeloma-specific therapy
* At least 4 weeks since participation in any clinical trial that involved an investigational drug or device
* No concurrent therapy with any of the following:

  * Corticosteroids (e.g., hydrocortisone, prednisone, prednisolone, dexamethasone [Decadron])

    * Inhaled steroids used for treatment of allergic rhinitis or pulmonary disease allowed
  * Thalidomide
  * Interferon
  * Growth factors, interleukins, or other cytokines (except filgrastim [G-CSF] as outlined in the protocol, or erythropoietin)
  * Cytotoxic chemotherapy agents (except cyclophosphamide for stem cell mobilization and high-dose melphalan)
  * Immunosuppressive drugs
  * Experimental therapies
  * Radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borrello, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Noonan KA, Huff CA, Davis J, Lemas MV, Fiorino S, Bitzan J, Ferguson A, Emerling A, Luznik L, Matsui W, Powell J, Fuchs E, Rosner GL, Epstein C, Rudraraju L, Ambinder RF, Jones RJ, Pardoll D, Borrello I. Adoptive transfer of activated marrow-infiltrating lymphocytes induces measurable antitumor immunity in the bone marrow in multiple myeloma. Sci Transl Med. 2015 May 20;7(288):288ra78. doi: 10.1126/scitranslmed.aaa7014. PMID 25995224

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was one screen failure.
Groups:
- MILs in Patients Undergoing an Autologous Peripheral SCT: therapeutic autologous lymphocytes
  therapeutic tumor infiltrating lymphocytes
  melphalan
  autologous hematopoietic stem cell transplantation
Period: Collection of MILs
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Relapsed | 1
Period: Generation of MILs Product
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Started | 23
Completed | 22
Not Completed | 1
Not completed — Relapsed | 1
Period: Administration of ASCT+MILs
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Started | 22
Completed | 4
Not Completed | 18
Not completed — Death | 10
Not completed — Lack of Efficacy | 8

BASELINE CHARACTERISTICS:
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 56 [30 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Hematopoietic Engraftment
Description: Days to absolute neutrophil count > 500 cells per microliter.
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: days
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
days | 17.9 [12 to 32]

2. Primary Outcome: Disease Response
Description: Percentage of participants with partial or complete response by Bladé criteria. Partial response is defined as a >= 50% decrease in serum paraprotein or 90% decrease in urinary light chains (for participants without measurable serum paraprotein). Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
Participants
  Complete Response | 7
  Partial Response | 6
  Stable Disease | 6
  Progressive Disease | 3

3. Primary Outcome: Feasibility of MILs Generation as Assessed by Percentage of Participants With Successful MIL Generation
Description: Success rate of expanding MILs in vitro and obtaining a protocol-specified product.
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
percentage of participants | 100

4. Secondary Outcome: T-cell Reconstitution as Determined by Absolute Lymphocyte Count (ALC)
Description: ALC counts trending over time.
Time Frame: Days 14, 28, 60, 180, and 360
Population: Data was not collected on one participant at the Day 28 and 180 timepoints, and data was not collected for eight participants at the Day 360 timepoint. Data was not collected on CD3+/CD4+/CD8+ cells for all participants.
Measure: Median (Full Range); unit: cells per microliter
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
cells per microliter
  Day 14 | 756 [105 to 2397]
  Day 28: number analyzed (Participants) | 21
  Day 28 | 1768 [349 to 3760]
  Day 60 | 1700 [530 to 3500]
  Day 180: number analyzed (Participants) | 21
  Day 180 | 1430 [650 to 2340]
  Day 360: number analyzed (Participants) | 14
  Day 360 | 1660 [690 to 2420]

5. Secondary Outcome: Survival
Description: Survival in months for participants who are alive (Overall Survival) and alive without disease progression (Progression-free survival). Disease progression is defined as a change from negative to positive on immunofixation or electrophoresis for participants previously in complete remission or a 25% increase in serum electrophoresis for participants not previously in complete remission. Partial response is defined as a >= 50% decrease in serum paraprotein or 90% decrease in urinary light chains (for participants without measurable serum paraprotein). Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
Time Frame: Up to 129 months
Measure: Median (Full Range); unit: months
Groups:
- MILs in Patients Undergoing an Autologous Peripheral SCT: therapeutic autologous lymphocytes
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
months
  Overall survival | 112.1 [39.9 to 128.7]
  Progression-free survival | 12.3 [8.8 to 69.03]

6. Secondary Outcome: Pneumococcal-specific Vaccine Responses
Description: CRM-197 Prevnar-specific vaccine responses that measure the T-cell response of the vaccine quantified as %CD3+/CFSE-low/IFN-gamma+.
Time Frame: At time of bone marrow harvest, Day 60 post-transplant, Day 180 post-transplant, and Day 360 post-transplant
Measure: Mean (Full Range); unit: %CD3+/CFSE-low/IFN-gamma+
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
%CD3+/CFSE-low/IFN-gamma+
  At time of bone marrow harvest | 21.5 [0.12 to 47.9]
  Day 60 post-transplant | 14.4 [0 to 38.2]
  Day 180 post-transplant | 23.4 [7 to 53]
  Day 360 post-transplant | 20.1 [0 to 49.7]

7. Secondary Outcome: Anti-tumor Immune Responses
Description: Myeloma lysate response that measures the T-cell response quantified as %CD3+/CFSE-low/IFN-gamma+.
Time Frame: At time of bone marrow harvest, Day 60 post-transplant, Day 180 post-transplant, and Day 360 post-transplant
Measure: Mean (Full Range); unit: %CD3+/CFSE-low/IFN-gamma+
Arm/Group | MILs in Patients Undergoing an Autologous Peripheral SCT
Number analyzed (Participants) | 22
%CD3+/CFSE-low/IFN-gamma+
  At time of bone marrow harvest | 1.58 [0 to 12.6]
  Day 60 post-transplant | 14.1 [0 to 44.3]
  Day 180 post-transplant | 18.1 [0.6 to 50.1]
  Day 360 post-transplant | 12.7 [0 to 31.8]

ADVERSE EVENTS:
Time Frame: Up to Day 360
Description: Per protocol, only adverse events (AEs) that were attributed to the study product (MILs) were collected and reported. AEs were collected daily through the date of engraftment, weekly through Day 28, and then at Days 60, 180, and 360.
Arm/Group | ASCT+MILs
All-Cause Mortality (participants affected / at risk) | 10/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASCT+MILs (N=22)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASCT+MILs (N=22)
Pain - abdomen (Musculoskeletal and connective tissue disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Blurred vision (Nervous system disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 9 (9)
Depression (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 17 (19)
Fever (Investigations) | 4 (4)
Headache (Nervous system disorders) | 7 (8)
Hypotension (Cardiac disorders) | 6 (6)
Insomnia (Nervous system disorders) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 2 (3)
Lightheadedness (Nervous system disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 9 (11)
Nausea (Gastrointestinal disorders) | 16 (18)
Neuropathy (Nervous system disorders) | 15 (21)
Neutropenic fever (Infections and infestations) | 5 (5)
Pain - calf (Musculoskeletal and connective tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 12 (22)
Sore throat (Skin and subcutaneous tissue disorders) | 7 (7)
Tachycardia (Cardiac disorders) | 3 (3)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes